CLINICAL TRIAL: NCT05331352
Title: Attachment Style and Mentalization Impact Among Women Victims of Domestic Violence
Acronym: FEMATAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: University of Franche-Comté (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020/546
Record Dates: First submitted 2021-10-04; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Violence, Domestic
Keywords: Domestic violence; Attachment; Mentalization; Victimization; Psychic elaboration of the trauma

STUDY DESIGN:
Intervention Model Description: First group : women following a psychotherapy Second group : women unfollowing a psychotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects following a psychotherapy (Experimental): Domestic violence victims following a psychotherapy 15 subjets Aged from 20 to 55
  Interventions: Behavioral: Semi-structured interviews; Behavioral: Projective methode; Behavioral: Selfreported
- Subjects unfollowing a psychotherapy (Experimental): Domestic violence victims unfollowing a psychotherapy 15 subjects Aged from 20 to 55
  Interventions: Behavioral: Semi-structured interviews; Behavioral: Projective methode; Behavioral: Selfreported

INTERVENTIONS:
Behavioral: Semi-structured interviews — Interview
Behavioral: Projective methode — Rorschach + thematic aperception test
Behavioral: Selfreported — RSQ - PBI - RFQ - QSCPGS - SSQ6 - ÉCHELLES DE CUNGI - STAI - PCL-S - IES-R

SUMMARY:
Attachment and mentalization with a population of domestic violence victims Domestic violence is one of the most common forms of domestic violence. Multiform and complex, it affects all backgrounds and all ages. According to a survey instituted by the government of Emmanuel Macron, 219,000 women were recognized as victims of domestic violence in 2017. This phenomenon is not without questioning the scientific scene. Also, this study focus on the quality of the attachment because if this bond is insecure, it can constitute a point of vulnerability in self-construction and impact on future relational modalities.

DETAILED DESCRIPTION:
The security of the bond of attachment depends on the capacity of the maternal figure, or her substitute, to understand and respond in an adapted and consistent manner to her baby. In addition, it has also been established that when disruptions occur in the security of attachment bond, the quality of mentalization is impacted. But, mentalization is the quality and quantity of psychic representations available to allow someone understanding and thinking about his links to others and to himself. This is an essential asset in the release of situations of violence and in overcoming trauma because it participates in psychic development. That's why this research focuses on early relationships and the quality of mentalization with a cohort of thirty women victims of domestic violence, consultant within the Legal Medicine department of the CHU of Besançon. This research focuses on two groups of subjects: women who managed to get out of violent relationship (15 subjects) and others who did not (15 subjects). The research methodology includes several tools: two projective tests (Rorschach and TAT), ten self-questionnaires (which assess attachment, stress, social support, relational quality with the main attachment figures, the image of the Self-body, quality of mentalization), a clinical research interview and presentation of the AAI. The observation of this population will highlight the impact of the early environment in the psychic construction of the subject and the victim's destiny. Moreover, this study will look at the role of psychotherapeutic follow-up in the quality of mentalization.

ELIGIBILITY:
Inclusion Criteria:

* Women over 20 years old, victims of domestic violence
* With european culture
* Separated from their abusive partner
* Consulting the Legal Medicine Department in Besançon University Hospital

Exclusion Criteria:

* Refusal to participate

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study entolls women suffering from domestic violence
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Security of the current attachment | Month 12
  Relationship Scale Questionary (RSQ)
  Description : 30 questions Answers : - 5 (not like me at all to) + 5 (very like me)
  Cotation :
  self-model scale : - 4 to + 4 model of others : - 4 to + 4 positive self-model and positive model of others = secure positive self-model and negative model of others = insecure detached negative self-model and positive model of others = insecure worried negative self-model and negative model of others = insecure fearful
Security of the early attachment | Month 12
  Adult Attachment Interview (AAI : Main, George & Kaplan, 1984 ; Pierrehumbert et al., 1999)
  Description : 20 questions Free answers
  Cotation : Edicode, Pierrehumbert Fluidity = 1 to 9 Coherence = 1 to 9 Reflexive = 1 to 9 Authentic = 1 to 9
  Scores have to be high
Mentalization | Month 12
  The Reflective Functioning Questionnaire (RFQ : Fonagy & al., 2016)
  The 8-item RFQ Reflective Functioning Questionnaire comprises two subscales each of 6 items (Uncertainty and Certainty about mental states) The two scales operate with a Likert scale of 7 points that evaluate the degree of agreement of the subject with the sentences presented in each item.
  The items of Uncertainty or RFQ_U correspond to statements such as "Often very strong feelings cloud my thinking", they are recorded to detect extreme levels of uncertainty about mental states, in the following way 0, 0, 0, 0, 1, 2, 3, so that high scores reflect hypomentalization.
  Scores have to be medium
  The items corresponding to Certainty of mental states or RFQ_C contemplate statements such as "When I get angry I say things without really knowing why I say them" which are recorded as 3, 2, 1, 0, 0, 0, 0, in such a way that a 6 low degree of agreement reflects Hypermentalization.
  Scores have to be medium
Quality of early relationship | Month 12
  Parental Bonding Instrument (G. Parker, H. Tupling and R.B. Brown) Two scales termed 'care' and 'overprotection' or 'control', measure fundamental parental styles as perceived by the child.
  25 item questions, including 12 'care' items and 13 'overprotection' items. Likert scale : "very like" (+3) or very dislike (-3).
  In addition to generating care and protection scores for each scale, parents can be effectively "assigned" to one of four quadrants:
  Mothers : care score = 27.0 / protection score = 13.5. Fathers :care score = 24.0 / protection score = 12.5. High care and high protection means "affectionate constraint". High protection and low care means "affectionless control". High care and low protection means "optimal parenting". Low care and low protection means "neglectful parenting".

SECONDARY OUTCOMES:
PTSD | Month 12
  Cungi's Scale 8 items Subject evaluates the importance for him of each of the items with a rating ranging from 1, very little impact at 6, extremely high impact. Score have to be low
  State-Trait Anxiety Inventory (STAI : Spielberg, 1983) Measures how the subject feels right now on 40 items with answer choices of 1 = not at all / almost never, 2 = somewhat/sometimes, 3 = moderately so / often, and 4 = very much so / almost always.
  Item scores are added to obtain subtest total scores. The score range for each subtest is 20-80, the higher score indicating anxiety. The cut point of 39-40 has been suggested to detect clinically significant symptoms.
  Impact of Event Scale Revisited (IES-R : Horowitz, Wilner, & Alvarez, 1979) 7 additional questions and a scoring range of 0 to 88. Scores that exceed 24 can be quite meaningful 33 and above : PTDS

OTHER OUTCOMES:
The social support | Month 12
  The social support questionnaire SSQ6 (Sarason et al., 1987) 6-item measure of social support. For each of the 6 items, respondents indicate the number of people available to provide support in each of 6 areas and then rate the overall level of satisfaction with the support given in each of the areas.
  For each item, the respondent makes a list of the people he can count on in the situation described (maximum 9 people) and expresses his degree of satisfaction (from 1 to 6) with this support.
  We then calculate two total scores, one of availability (N=number of people cited) and the other satisfaction (S), which correspond respectively to the sum of the "number" (N score) and "satisfaction" (S score) scores obtained in each of the six items.
  N score varies from 0 to 54 and the S score from 6 to 36. Both scores must be as high as possible
The self-satisfaction | Month 12
  The self-satisfaction with the body satisfaction and global self-perception questionnaire (QSCPGS) Total score ranges from -100 to +100, each of the 20 items ranging from -5 to +5.
  The sign of value surrounded is a function of the proposal he has chosen to define himself.
  The sum of the 20 values gives the total score. If three or more answers lack, the QSCPGS is not valid.
  For quality analysis, the calculation of the number of hits, negative replies and neutral gives an indication of the perception that the subject of himself. This value is given as a percentage positive, negative and neutral. An item analysis by item, as well as the total and both factors can be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Houari Maïdi, PhD, Study Director — Université de Bourgogne Franche-Comté
Locations (1):
- CHU Besançon, Besançon, Bourgogne-Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cesari J, Belot RA, Thomas C, Jollivet M, Martin E, Clesse C. Affect regulation, mentalization, and attachment in intimate partner violence survivor women: A quasi-experimental controlled trial. Psychol Trauma. 2025 Oct 30. doi: 10.1037/tra0002047. Online ahead of print. PMID 41166191